CLINICAL TRIAL: NCT03294824
Title: Study of Natural Killer Immunity During Infections With CMV or AdV After Allogeneic Hematopoietic Stem Cells
Brief Title: Non Randomized Comparative Study With Control
Acronym: Allo-NK-CMV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P111107; IDRCB (Other: 2013-A00825-40)
Record Dates: First submitted 2016-02-15; First posted 2017-09-27 (Actual); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Allogeneic Hematopoietic Stem Cell Transplantation
Keywords: NK cells; Cytomegalovirus; adenovirus; Allogeneic transplantation
MeSH Terms: conditions — Adenoviridae Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- patients who reactivate CMV or AdV after allogeneic HSCT: allotransplanted patients who reactivated respectively CMV (n=30) and AdV (n=10)
  Interventions: Other: blood sample
- Control group: allogeneic HSC transplanted patients: allotransplanted patients who didn't reactivate CMV
  Interventions: Other: blood sample
- Healthy donors group: healthy donors serologically + for CMV
  Interventions: Other: blood sample

INTERVENTIONS:
Other: blood sample — peripheral blood samples are collected

SUMMARY:
NK cells are lymphocytes who play a role in the control of viral infections , tumor and fœtal tolerance. They belong to innate immune cells but they have a link with adaptative immunity. Indeed, after some viral infections such as CMV, Chikungunya, B hepatitis etc, a subset of NKG2C+ NK cells expands and can transfer, in murine models, a " memory " that can better control CMV infections. CMV reactivation is a major cause of morbidity and mortality after allogeneic hematopoietic ste cell transplantation in humans. The aim of this prospective study is to evaluate the role of NK cells, in particular NKG2C+ NK cells in the control of CMV but also Adenovirus after allo HSCT. Peripheral NK cells from 30 and 10 patients who reactivated respectively CMV and AdV are prospectively studied (extensive phenotyping and functional studies before and after administration of anti viral drugs) and compared with 30 allotransplanted patients who didn't reactivate CMV in a pair analysis, and 30 healthy donors serologically + for CMV.

DETAILED DESCRIPTION:
For both groups: 28ml of peripheral blood samples are collected at different points. Group 1 : before and after anti viral treatment . Control group 2: one point after allo-HSCT; Control group 3: 1 point before transplant. Phenotypical study of NK cells: activating and inhibitory receptors, activation and differentiation's markers. Phenotypical studies of the ligands on infected cells. Genotypic study of KIR receptors (Kirotype); functional studies: polyfunctionality essay (flow cytometry): degranulation CD107a, IFNg, TNFa production).

ELIGIBILITY:
Inclusion Criteria:

1. patients who reactivate CMV or AdV after allogeneic HSCT ;

   * Age>18 years; indication for a antiviral treatment:
   * at least 1 PCR CMV>1000 copies/ml or 1 PCR ADV>1000 copies/ml or at least 2 ADV PCR positive - sites (stools, throat, urines);
   * signed informed consent;
2. Control group: allogeneic HSC transplanted patients;

   * Age>18 years; no CMV or AdV reactivation ;
   * signed informed consent;
3. Healthy donors group: HSC donor;

   * Age>18 years;
   * signed informed consent

Exclusion Criteria:

none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Allogeneic HSCT for malignant or non malignant hematological disease in adult patients
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2013-09-27 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Nk cells phenotype (activation, differentiation, memory NK cell) and function (cytoxicity and cytokines production) measured by flow cytometry | Change from "before antiviral treatment", " half treatment" (1 week or 2 week after the beginning of the treatment), 1 month "post treatment" and 3 month "post treatment"
  CD3-CD56+ NK cells will be analyzed by Flow cytometry with an appropriate monoclonal antibodies (mAb) cocktail: anti-CD3 ,CD56, CD16, CD159a/NKG2A , CD85J; HLA-DR ; CD62L , CD161; KIR2DL1 and KIR3DL1, and KIR2DL2/KIR2DL3.
  The state of NK cells differentiation and maturation will be assessed by the analyze of thoses phenotypic markers and will be compared with healthy donors.
NK cells cytoxicity and cytokines production when incubated with standard HLA class I negative K562 target cells | Change from "before antiviral treatment", " half treatment" (1 week or 2 week after the beginning of the treatment), 1 month "post treatment" and 3 month "post treatment"
  Polyfunctional assay will test the capacity of NK cells degranulation and production of cytokines when incubated with standard HLA class I negative K562 target cells in the presence of anti-CD107a ,IFN-g, or TNF-a mAb.
  The state of NK cells differentiation and maturation will be assessed by the analyze of thoses phenotypic and will be compared with healthy donors.

SECONDARY OUTCOMES:
Effect of CMV and AdV infection compared with healthy donors | Change from "before antiviral treatment", " half treatment" (1 week or 2 week after the beginning of the treatment), 1 month "post treatment" and 3 month "post treatment"
  The state of NK cells differentiation and maturation will be assessed by the analyze of thoses phenotypic and functional markers and will be compared with healthy donors.
In vitro Nk cells ligands analyzes on infected cells by CMV | approximately 18 months after Study Completion Date (last participant's last visit)
  Monocyte are differentiated in macrophage cells and infected by the CMV strain TB40/E. Nk cell ligands will be analyzed on infected cells. NK cells from infected patients post allogenic transplantation will be tested against in vitro infected cells.
  Being a model in vitro, it is not possible to determine in advance which ligands will be identified.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Nguyen Quoc, Doctor, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Pitié Salpêtriere, Paris, France

IPD SHARING:
Plan to Share IPD: No